CLINICAL TRIAL: NCT00741299
Title: Association Between Tobacco Smoking and Bipolar Affective Disorder.Clinico-epidemiological, Cross-sectional, Retrospective Study.
Brief Title: A Study of the Association Between Tobacco Smoking and Bipolar Affective Disorder
Status: Completed | Type: Observational
Sponsor: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Anatoly Dr. Kreinin, Director of psychiatric department, Tirat Carmel Mental Health Center
Other Study IDs: GKN2007; GKN2007
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Bipolar Disorder
Keywords: bipolar affective disorder, Smoking
MeSH Terms: conditions — Bipolar Disorder; Smoking

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine whether tobacco smoking is associated with bipolar affective disorder (severity of depressive and manic symptoms, presence of psychotic symptoms, history of a suicide attempts and other clinical features.)

DETAILED DESCRIPTION:
An association exists between smoking and schizophrenia, independent of other factors and related to psychotic symptomatology. Only a few small descriptive studies have examined the prevalence and correlates of tobacco use among bipolar patients with conflicting results. Patients who smoke score higher on rating scales for psychotic symptoms than their non-smoking peers. While the association of smoking with psychotic symptomatology in schizophrenia is established, such association according to bipolar affective disorder has been reported in a few studies and remains unclear. Also a few studies reported about association of smoking with depressive and manic symptoms, and with suicidal behavior in bipolar patients. Thus further investigation of these issues is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 male or female
* DSM -IV criteria for bipolar I affective disorder
* Ability and willingness to sign informed consent for participation in the study

Exclusion Criteria:

* Unwillingness or inability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will consist of all patients ascertained in database of Tirat Carmel Mental Health Center and Psychiatric Outpatients Clinic, Rambam Medical Center
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Relationship between smoking and other factors including: bipolar subtype, current and past clinical status, illness severity,history of a suicide attempts, age of bipolar onset, gender, education, social class, economic status. | One interview session

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Kreinin, MD, PHD, Principal Investigator — B. Rappaport Faculty of Medicine, Technion, Haifa
Locations (1):
- Tirat Carmel Mental Health Center, Tirat HaCarmel, Tirat HaCarmel, Israel

REFERENCES:
- [Derived] Kreinin A, Novitski D, Rabinowitz D, Weizman A, Grinshpoon A. Association between tobacco smoking and bipolar affective disorder: clinical, epidemiological, cross-sectional, retrospective study in outpatients. Compr Psychiatry. 2012 Apr;53(3):269-74. doi: 10.1016/j.comppsych.2011.04.063. Epub 2011 Jun 12. PMID 21664608